CLINICAL TRIAL: NCT04401072
Title: Survey Studying the Change in the Attitude and Behaviour of the Egyptian Population Toward COVID 19 Pandemic During the Holy Month Ramadan .
Brief Title: Attitude of Egyptian Population Toward COVID 19 in Ramadan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Other Study IDs: covid 19 in ramadan
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Covid 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the COVID 19 pandemic and after new cases started to appear in Egypt in march 2020 the Egyptian government issued movement restrictions and placed areas into quarantine to reduce the spread of the virus. Egyptian citizens were encouraged to adopt personal protective measures, such as staying at home , increasing personal hygiene and wearing protective face masks. Ramadan is a holy month and a very special event for all the Muslims worldwide including the Egyptian Muslims . the Egyptians have many rituals and traditions special for Ramadan . normally Egyptian people tend to go to family gatherings and go out for iftar and suhoor in Ramadan .the markets also tend to be very crowded and full of people in Ramadan for buying food and other preparations for Ramadan and Eid Al Fitr. This all can lead to crowdingof people in the streets and markets and increases the chance of the spread of the virus and the chance of infection.Public Awareness play a major rule in reducing the spread of COVID 19 so in this study a survey is done to measure the attitude of the Egyptian population toward COVID 19 in Ramadan and to evaluate if the rituals and traditions in the holy month are affecting the spread of COVID 19 in Egypt.

DETAILED DESCRIPTION:
The survey will enroll as many individuals of the Egyptian population as possible in the survey portion of the study - The number of participates have no limitations, at least 500 participants.

The survey will be enrolled in online google form, face to face interview(this will be reduced to encourage social isolation) & semi-structured telephone interviews if possible.

The research procedures:

An online survey link will include questions regarding the attitude and behaviour of the Egyptian population during the COVID-19 outbreak in Ramadan and to evaluate if people are practicing their normal rituals and traditions in the holy month and how can this affect the COVID 19 spread in Egypt.

Face to face and semi-structured interviews if possible: For those Egyptian citizens who state that they would like to participate in an interview, a random sample will be contacted.

Inclusion Criteria:

Egyptian population of any age group

Exclusion Criteria:

none

ELIGIBILITY:
Inclusion Criteria:

Egyptian population

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian population of all age groups
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Attitude of the Egyptian population during the COVID 19 pandemic in Ramadan | 6 months
  evaluate theattitude and behaviour and of the Egyptian population during COVID 19 pandemic in Ramadan

CONTACTS AND LOCATIONS:
Locations (1):
- Damanhour University, Damanhur, Beheira, Egypt

IPD SHARING:
Plan to Share IPD: Undecided